CLINICAL TRIAL: NCT07302620
Title: HEPARINS: INTERFERENCE IN ARGATROBAN MEASUREMENT
Acronym: HIMA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9457
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Thromboembolic Disease
Keywords: Thromboembolic Disease; HEPARINS; ARGATROBAN; Unfractionated heparin (UFH); Low molecular weight heparins (LMWH); Anti-Xa and anti-IIa activity
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Unfractionated heparin (UFH) and low molecular weight heparins (LMWH) provide anticoagulation through their anti-Xa and anti-IIa activity. This anti-IIa activity can lead to an overestimation of argatroban's activity when switching to an anti-IIa anticoagulant such as argatroban. This situation can be critical because argatroban is generally administered following heparin therapy due to suspected heparin-induced thrombocytopenia. Therefore, there is both a significant thrombotic risk induced by the underlying condition and a hemorrhagic risk induced by the anticoagulation. For this reason, it is important to be able to accurately monitor the anti-IIa activity of argatroban. To date, the test used to determine the anti-IIa activity of argatroban at the Hematology Laboratory of the Strasbourg University Hospitals (HUS) is a modified thrombin time (with a calibration curve adapted for argatroban). When switching between several molecules with anti-IIa activity, this test does not allow for the differentiation of the anti-IIa activity attributable to each anticoagulant.

There are no data in the literature to determine whether heparins interfere with this test, and if so, its extent.

ELIGIBILITY:
Inclusion Criterias:

* Adult patient (≥ 18 years)
* Patient anticoagulated with UFH or LMWH
* Sample sent to the Hematology Laboratory of the University Hospitals of Strasbourg (HUS) and analyzed for measurement of the anti-Xa activity of an anticoagulant in routine care

Exclusion Criteria:

* Patient receiving an anticoagulant other than UFH or LMWH
* Insufficient sample volume

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥ 18 years) anticoagulated with UFH or LMWH
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pearson or Spearman correlation test | 1 hour after analysis
  * A correlation test (Spearman or Pearson) will be performed to compare anti-Xa activity with anti-IIa activity to determine if there is a significant correlation that could lead to an overestimation of argatroban's anti-IIa activity during a heparin-argatroban switch.
  * Spearman correlation uses the rank of the data to measure monotonicity between ordinal or continuous variables. Pearson correlation, on the other hand, detects linear relationships between quantitative variables with data following a normal distribution.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie - Unité d'Hémostase - CHU de Strasbourg - France, Strasbourg, France